CLINICAL TRIAL: NCT06135454
Title: Open Wedge High Tibial Osteotomy Versus Double Level Osteotomy
Brief Title: Comparison of Outcomes Between Open Wedge High Tibial Osteotomy and Double Level Osteotomy in Antromedial Knee Arthritis With Extra Articular Deformity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd Elgawad Mohamed Abd Elgawad Ahmed, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Knee Osteoarthritis
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Wedge High Tibial Osteotomy (Experimental)
  Interventions: Procedure: Open Wedge High Tibial Osteotomy
- Double Level Osteotomy (Experimental)
  Interventions: Procedure: Open Wedge High Tibial Osteotomy; Procedure: Double Level Osteotomy

INTERVENTIONS:
Procedure: Open Wedge High Tibial Osteotomy — For OWHTO,The osteotomy plane, directed from 30 to 35 mm distal to the medial tibial plateau to 10-15 mm distal to the lateral tibial plateau in the coronal plane, was marked by two Kirschner wires with threaded tips. A transverse osteotomy was performed, leaving the lateral cortex intact as a hinge. After the ascending osteotomy and opening. The medial opening gap was filled with two β-TCP wedges and fixed with a TomoFix anatomical plate and locking screws .
Procedure: Double Level Osteotomy — The DLO was started from a lateral DFO. A 5-6-cm incision was made proximally at the distal femur from the lateral femoral epicondyle.Two Kirschner wires with threaded tips were inserted to make a length between the wires that was preoperatively planned as the lateral closed osteotomy. Transverse and ascending osteotomies were performed using a Precision Oscillating Tip Saw. The gap was closed and fixed using a TomoFix medial distal femur anatomical plate , which was bent for the lateral distal femur. The subsequent OWHTO was performed as described above.
  Arms: Double Level Osteotomy

SUMMARY:
To compare the radiographic and clinical outcomes of varus osteoarthritic knees treated with an open-wedge high tibial osteotomy (OWHTO) alone or with a double-level osteotomy (DLO). It was hypothesized that treatment with DLO would prevent the joint line obliquity (JLO) , optimize post-operative limb alignment and provide better clinical and radiological outcomes after surgery than medial opening-wedge high tibial osteotomy (OWHTO) alone for patients with medial compartment osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease characterized by erosion of the articular cartilage, hypertrophy of the bone at the margins and subchondral sclerosis(1). Osteoarthritis of the knee is a common problem causing significant knee pain and disability. Medial compartment osteoarthritis is predisposed to be varus deformity of the knee(2). High tibial osteotomy (HTO) is a well-established method for treatment of medial Uni compartmental-knee osteoarthritis and correction of varus deformity(3).Double level osteotomy recently used as another method for treatment this problem to improve outcomes and decrease complication(4).

ELIGIBILITY:
Inclusion Criteria:

* Patients that are indicated for surgery for medial compartment osteoarthritis only (medial joint line tenderness, varus tibiofemoral malalignment) with classification of Kellgren Lawrence grade (1/2/3)
* Age between 40 _ 60 years
* No associated bony fractures or deformities
* No associated ligamentous functional instability
* Varus more than or equal 15 degrees

Exclusion Criteria:

* Age younger than 40 or older than 60 years
* Secondary Arthritis (Inflammatory arthritis, post-traumatic osteoarthritis, active knee infection)
* Lateral Compartment OA or patellofemoral OA

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of joint line obliquity (JLO) in the two groups. | Preoperative , three months postoperative , one year postoperative
  Postoperative limb alignment using bilateral standing anteroposterior full-length views of both lower limbs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akamatsu Y, Nejima S, Tsuji M, Kobayashi H, Muramatsu S. Joint line obliquity was maintained after double-level osteotomy, but was increased after open-wedge high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2022 Feb;30(2):688-697. doi: 10.1007/s00167-020-06430-6. Epub 2021 Jan 12. PMID 33433634
- [Background] Babis GC, An KN, Chao EY, Rand JA, Sim FH. Double level osteotomy of the knee: a method to retain joint-line obliquity. Clinical results. J Bone Joint Surg Am. 2002 Aug;84(8):1380-8. doi: 10.2106/00004623-200208000-00013. PMID 12177268
- [Background] Schuster P, Rathgeb F, Mayer P, Michalski S, Hielscher L, Buchholz J, Kruger L, Richter J. Double level osteotomy for medial osteoarthritis and bifocal varus malalignment has excellent short-term results while maintaining physiologic radiographic joint parameters. Knee Surg Sports Traumatol Arthrosc. 2023 Aug;31(8):3124-3132. doi: 10.1007/s00167-022-07247-1. Epub 2022 Dec 10. PMID 36494478